CLINICAL TRIAL: NCT07232069
Title: Prospective RandomizEd Evaluation and Management of Premature aTherosclerosis
Brief Title: PRE-EMPT: Prospective RandomizEd Evaluation and Management of Premature aTherosclerosis
Acronym: PRE-EMPT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of North Carolina, Chapel Hill (Other); Massachusetts General Hospital (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00118744; UG3HL181434 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease Risk Factors Multiple; Coronary Artery Disease Progression; Prevention & Control; Premature Atherosclerosis
Keywords: Prevention; Heart Disease Prevention; Family History of Heart Disease; At risk for heart disease; coronary artery calcium; non-calcified coronary plaque
MeSH Terms: interventions — Rosuvastatin Calcium; Tablets; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- rosuvastatin 20mg plus colchicine-matched placebo (Experimental): statin plus placebo (two pills once daily)
  Interventions: Drug: Rosuvastatin 20 Mg Oral Tablet; Drug: Placebo
- colchicine 0.5mg plus rosuvastatin-matched placebo (Experimental): anti-inflammatory plus placebo (two pills once daily)
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet Once Daily; Drug: Placebo
- rosuvastatin 20mg plus colchicine 0.5mg (Experimental): statin plus anti-inflammatory (two pills once daily)
  Interventions: Drug: Rosuvastatin 20 Mg Oral Tablet; Drug: Colchicine 0.5 MG Oral Tablet Once Daily
- placebo plus placebo (Placebo Comparator): Placebo and placebo (two pills once daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin 20 Mg Oral Tablet — Statin
  Other Names: Crestor
  Arms: rosuvastatin 20mg plus colchicine 0.5mg; rosuvastatin 20mg plus colchicine-matched placebo
Drug: Colchicine 0.5 MG Oral Tablet Once Daily — Anti-inflammatory
  Other Names: Lodoco
  Arms: colchicine 0.5mg plus rosuvastatin-matched placebo; rosuvastatin 20mg plus colchicine 0.5mg
Drug: Placebo — Placebo, non-active, drug-matched
  Arms: colchicine 0.5mg plus rosuvastatin-matched placebo; placebo plus placebo; rosuvastatin 20mg plus colchicine-matched placebo

SUMMARY:
Heart disease is the leading cause of death for men, women, and people of most racial and ethnic groups in the United States. This clinical trial will test if screening and early treatment of mild heart disease works.

PRE-EMPT will screen individuals at low 10-year risk of heart disease with heart disease risk factors to identify those who already have early cholesterol build up, also called "plaque", in their heart arteries. It consists of two phases:

1. A Screening Study - Participants will be assessed for plaque by one or both of these scans.

   * Coronary Artery Calcium (CAC) Scan: A CT scan that looks for calcium or plaque in heart arteries.
   * Coronary CT Angiography (CCTA) Scan: A CT scan that uses contrast dye to create detailed 3D pictures of heart arteries to look for plaque.
2. A Treatment Trial (approximately 1,500 participants) - Based on the results of the CCTA, participants may be randomized into a two-year trial to test medications aimed at reducing or stabilizing plaque. Participants will have a 1 in 4 chance of receiving only placebo, and a 3 in 4 chance of receiving at least one active medication. Participants will take two pills once a day-either both active medications, one active and one placebo, or both placebos.

   * Rosuvastatin 20 mg: a cholesterol-lowering medicine
   * Colchicine 0.5 mg: a medication that lowers inflammation

Everyone in the trial will be given information and advice on heart-healthy diet and lifestyle.

Participants will have up to two in-person visits for the screening study, then phone visits for the Treatment Trial at the beginning, 3 months, 12 months and 24 months when they will also have an in-person visit for a CCTA Scan. Participants will have blood drawn using an at-home collection device mailed to their home at the beginning, 3 months, and end of the study.

DETAILED DESCRIPTION:
The PRE-EMPT trial will be a 2x2 factorial, double-masked, placebo-controlled randomized trial of the effects of high-intensity statin and low-dose colchicine, alone and in combination, on CCTA-defined Non-Calcified Coronary Plaque (NCCP) volume at 2 years. Participants found through the screening study with CAC 1-99, or through the known plaque pathway, will be eligible for the trial if they have NCCP without severe stenosis or any other exclusion criteria. Study drug will be delivered directly to participants' homes, lab samples will be self-collected at home, and all study visits will be virtual except the imaging visits (up to 3 over 2 years). The only in-person study activities will be the CAC scan, if applicable, and CCTA at baseline and 2 years. The investigators anticipate that this approach will be attractive to middle-aged, busy individuals who are otherwise healthy and asymptomatic. Importantly, all participants in PRE-EMPT will receive an mHealth lifestyle intervention designed to support behavioral modification, ensuring that all individuals benefit from evidence-based strategies for cardiovascular risk reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 40-60 years; Men aged 30-50 years
2. Willing and able to provide informed consent and comply with study procedures
3. Smart phone user
4. Use of highly effective contraception by females with reproductive potential.
5. CAC score 1-99 in the screening study or entry through the known plaque pathway (with mild CAC or CAC<100 if known; elevated CAC on baseline CCTA is not exclusionary in the known plaque arm)
6. Diagnostic baseline CCTA with NCPV ≥10 mm3 as assessed by the central core lab

Exclusion Criteria:

1. Clinical diagnosis of ASCVD Diagnosis (MI, stroke, arterial revascularization) or current symptoms thought to be from coronary artery disease
2. PREVENT ASCVD 10-year risk ≥5% (if known)
3. Diabetes Mellitus (DM) as defined by any of the following: new DM diagnosis in the medical record or HbA1C of 6.5% or greater. (if known)
4. LDL-C ≥190mg/dL (most recent, if known)
5. HIV (if known)
6. Severe liver disease or untreated Hepatitis C infection (if known)
7. Pregnancy, lactation or intending to become pregnant during the study period of 2 years
8. eGFR <45mL/min/1.73m2 (if known)
9. AST or ALT >1.5x the upper limit of normal (if known)
10. BMI>40kg/m2
11. Allergy to iodinated intravenous contrast or other contraindication to CCTA
12. Current or previous use of lipid lowering therapy or colchicine
13. Known allergic reactions or sensitivity to the study intervention(s), including known intolerance or contraindication(s) to statin or colchicine, or long-term use of medications that are contraindicated with colchicine or rosuvastatin.
14. Systemic cancer undergoing active treatment
15. PREVENT ASCVD 10-year risk ≥5%
16. eGFR <45 ml/min/1.73m2 per baseline labs
17. Hemoglobin A1c ≥6.5% per baseline labs
18. LDL-C ≥190mg/dL per baseline labs
19. Severe proximal coronary artery stenosis as determined by the central core lab
20. Known contraindication to follow-up CCTA (e.g., new IV contrast allergy discovered during the baseline CCTA)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged 40-60 years old, Men aged 30-50 years old
Enrollment: 1500 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Non-calcified plaque volume (NCPV) on CCTA at 2 years, adjusted for baseline NCPV. | 2 years
  Plaque volume in mm3 in each group

SECONDARY OUTCOMES:
Number of participants with Drug Discontinuation | Up to 2 years
  Drug Tolerability outcome
Overall drug treatment adherence | Up to 2 years
  Number of days on study drugs
Safety events of special interest | Up to 2 years
  Number of safety events of special interest per group
Total plaque volume | Up to 2 years
  Plaque volume in mm3 per group
Low-attenuation plaque volume | Up to 2 years
  Low attenuated plaque volume in mm3 per group
Calcified plaque volume | Up to 2 years
  Calcified plaque volume in mm3 per group
Number of participants with stenosis | Up to 2 years
  Number of participants with stenosis per group
Segment involvement score | Up to 2 years
  Average score per group
Number of participants with qualitative calcified, partially calcified and non-calcified plaque composition | Up to 2 years
  Number of participants with each plaque composition description per group
Number of participants with High-risk plaque features (positive remodeling, spotty calcium, napkin ring sign) | Up to 2 years
  Number of participants with each plaque feature (high-risk) per group
Change in LDL-C (low-density lipoprotein cholesterol) | Baseline to 2 years
Change in non-HDL-C (high-density lipoprotein cholesterol) | Baseline to 2 years

IPD SHARING:
Plan to Share IPD: No